CLINICAL TRIAL: NCT01155284
Title: Combination Therapy With Sitagliptin (DPP 4 Inhibitor) and Lansoprazole (PPI) Inhibitor) to Restore Pancreatic Beta Cell Function in Recent-Onset Type 1 Diabetes
Brief Title: Combination Therapy With Sitagliptin and Lansoprazole to Restore Pancreatic Beta Cell Function in Recent-Onset Type 1 Diabetes
Acronym: REPAIR-T1D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanford Health (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Kurt Griffin, Principal Investigator, Sanford Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REPAIR-T1D
Record Dates: First submitted 2010-06-03; First posted 2010-07-01 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-08

CONDITIONS: Type 1 Diabetes
Keywords: diabetes; HGB A1C; Beta Cell Regeneration
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Sitagliptin Phosphate; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin and Lansoprazole (Experimental): Sitagliptin 50mg co-administered with Lansoprazole 30mg. Subjects age 11-17 years at Visit 2 will take 1 capsule of each once daily Subjects age 18-45 years at Visit 2 will take 2 capsules of each once daily
  Interventions: Drug: Sitagliptin and Lansoprazole
- Placebo (Placebo Comparator): Sitagliptin Placebo and Lansoprazole placebo capsules will be administered. Subjects age 11-17 years at Visit 2 will take 1 placebo capsule of each once daily Subjects age 18-45 years at Visit 2 will take 2 placebo capsules of each once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin and Lansoprazole — Sitagliptin (dispensed as 50 mg capsules)and Lansoprazole(dispensed as 30 mg capsules) or matching placebo
  * Subjects age 11-17 years at Visit 2 will take 1 capsule once daily
  * Subjects age 18-45 years at Visit 2 will take 2 capsules once daily
  Other Names: Januvia; Prevacid
  Arms: Sitagliptin and Lansoprazole
Drug: Placebo — Sitagliptin 50mg and Lansoprazole 30 mg or matching placebo will be given daily for 12 months. Subjects age 11-17 at visit 2 will take 1 capsule daily; age 18-45 will take 2 capsules daily.
  Other Names: Januvia; Prevacid
  Arms: Placebo

SUMMARY:
Sanford Research/USD proposes to study the combination therapy of oral administration of sitagliptin and lansoprazole versus placebo for the preservation of pancreatic beta cells still present in patients with recent-onset diabetes and possibly regenerating their beta cells, while safely down-regulating the autoimmune response directed against the beta cells.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes, based on American Diabetes Association criteria, recently diagnosed (within the 6 months before Screening) and confirmed by the presence of at least 1 diabetes related autoantibody (either glutamic acid decarboxylase [GAD], insulinoma-associated protein [IA 2], or insulin, the latter measured within 10 days after starting insulin therapy).
* Male or female aged between 11 and 45 years, inclusive.
* Able to swallow study capsules.
* Willing to comply with "intensive diabetes management" as directed by the investigator, with the goal of maintaining blood glucose as close to American Diabetes Association recommendations as possible.
* Willing to comply with the schedule of study visits and protocol requirements.

Exclusion Criteria:

* Use of a GLP 1R agonist or DPP 4 inhibitor within 1 month before enrollment.
* Use of a PPI within 1 month before enrollment.
* Use of an oral hypoglycemic agent within 1 month before enrollment or use of thiazolidinediones within 3 months before enrollment (although thiazolidinediones may be used <7days before enrollment).
* Females of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period.
* Females who are pregnant or breastfeeding at the time of enrollment.
* Subjects with any of the following conditions:

  * Renal insufficiency, defined as estimated glomerular filtration rate (GFR) less than 50 mL/min at Screening, calculated using the Modification of Diet in Renal Disease (MDRD) equation.
  * History of a serious hypersensitivity reaction to sitagliptin or lansoprazole, such as anaphylaxis or angioedema.
  * Severe hepatic insufficiency.
  * History of pancreatitis or gallbladder disease
  * Any significant medical condition, which in the opinion of the investigator or medical monitor would interfere with study participation.

Ages: 11 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2010-08; Primary Completion 2014-05 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Rabinovitch, MD, Principal Investigator — Sanford Research/USD; Diane L Hahn, LPN, Study Director — Sanford Research/USD
Locations (3):
- United States (3):
  - Rady Children's Hospital, San Diego, California
  - Children's - St. Paul, Saint Paul, Minnesota
  - Sanford Research/USD, Sioux Falls, South Dakota

REFERENCES:
- [Result] Griffin KJ, Thompson PA, Gottschalk M, Kyllo JH, Rabinovitch A. Combination therapy with sitagliptin and lansoprazole in patients with recent-onset type 1 diabetes (REPAIR-T1D): 12-month results of a multicentre, randomised, placebo-controlled, phase 2 trial. Lancet Diabetes Endocrinol. 2014 Sep;2(9):710-8. doi: 10.1016/S2213-8587(14)70115-9. Epub 2014 Jul 2. PMID 24997559

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four centers screened 79 participants were screened between August 2010 and May 2012. Participants aged 11-36 years, diagnosed with type 1 diabetes within the past 6 months were recruited. 9 participants were not randomized as 7 were deemed ineligible and 2 were lost to follow-up.
Pre-assignment Details: At a screening visit, participants underwent procedures to establish that all inclusion criteria were met and none of the exclusion criteria were met. All participants and if applicable, guardians provided written informed consent/assent at screening.
Groups:
- Sitagliptin and Lansoprazole: Oral Sitagliptin (100 mg for those age 18 -45 years, 50 mg for those age 11-17 years) and Lansoprazole (60 mg for those 18-45 years, 30 mg for those age 11-17 years for 12 months. Participants were then followed for an additional 12 months.
- Placebo: Placebo: Matching placebo was given daily for 12 months.
Period: Overall Study
Arm/Group | Sitagliptin and Lansoprazole | Placebo
Started | 47 | 23
Completed | 40 | 18
Not Completed | 7 | 5
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: 70 participants were randomized. After randomization, 2 participants withdrew (one was from treatment group and one from placebo group) before taking any drugs, leaving 46 participants in the active treatment group and 22 in the placebo.
Groups:
- Placebo: Matching placebo will be given daily for 12 months. Participants were then followed for an additional 12 months.
- Total: Total of all reporting groups
Arm/Group | Sitagliptin and Lansoprazole | Placebo | Total
Number analyzed (Participants) | 46 | 22 | 68
Age, Customized [Mean (Standard Deviation); unit: years]
  Age (years) | 15.5 (5.1) | 17.6 (6.9) | 16.2 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 10 | 29
  Male | 27 | 12 | 39
Days Post diagnosis [Mean (Standard Deviation); unit: Days] | 102.8 (51.8) | 104.7 (52.8) | 103.4 (51.7)
GAD antibody positive [Number; unit: participants] | 42 | 22 | 64
HLA DR Allele - Neither DR3 nor DR4 [Number; unit: participants] | 2 | 3 | 5
HLA DR Allele - DR3 only [Number; unit: participants] | 11 | 7 | 18
HLA DR4 Allele only [Number; unit: participants] | 19 | 6 | 25
HLA DR Allele - Both DR3 and DR4 [Number; unit: participants] | 14 | 6 | 20
Insulin use (units/kg per day) [Mean (Standard Deviation); unit: units/kg per day] | 0.43 (0.22) | 0.38 (0.17) | 0.41 (0.20)
2 -hour C-peptide Area Under Curve Result in Response to Standardized Mixed Meal Tolerance Test [Mean (Standard Deviation); unit: pmol/L] — C-peptide reflects how much insulin pancreatic beta cells are making. The MMTT measures how much insulin can be made. Blood samples for C-peptide were collected at baseline, 15, 30, 60, 90 and 120 minutes post-meal. Results are presented as the time weighted average concentration. To maintain consistency with prior reports, this has been labeled as "AUC," although it may be more accurate to describe this as an AUC mean (pmol/L), [true AUC (pmol*min/L) / 120 minutes]. Larger numbers are better, reflecting preservation of insulin production.
  pmol/L | 656 (385) | 747 (468) | 686 (413)
Glucose (mmol/L) [Mean (Standard Deviation); unit: mmol/L] — time weighed mean during mixed meal test
  mmol/L | 10.61 (3.35) | 10.47 (3.43) | 10.56 (3.35)
HbA1c (%) [Mean (Standard Deviation); unit: %] | 7.19 (1.09) | 7.15 (1.13) | 7.18 (1.09)
IDA-HbA1c (%) [Mean (Standard Deviation); unit: %] | 8.9 (1.53) | 8.68 (1.43) | 8.83 (1.49)

OUTCOME MEASURES:

1. Primary Outcome: 2 Hour C-peptide AUC in Response to MMTT
Description: Blood samples for C-peptide were collected at baseline (pre-meal) and 15, 30, 60, 90 and 120 minutes post-meal.
Time Frame: Month 12
Population: Of the 70 subjects randomized, 58 completed treatment and analysis.
Measure: Median (95% Confidence Interval); unit: pmol/L
Groups:
- Sitagliptin and Lansoprazole: Sitagliptin and Lansoprazole: Sitagliptin (dispensed as 50 mg capsules)and Lansoprazole(dispensed as 30 mg capsules) given daily for 12 months.
  * Subjects age 11-17 years at Visit 2 will take 1 capsule once daily
  * Subjects age 18-45 years at Visit 2 will take 2 capsules once daily
- Placebo: Matching placebo will be given daily for 12 months. Subjects age 11-17 at visit 2 will take 1 capsule daily; age 18-45 will take 2 capsules daily.
Arm/Group | Sitagliptin and Lansoprazole | Placebo
Number analyzed (Participants) | 40 | 18
pmol/L | 358 [308 to 563] | 495 [299 to 675]
Statistical Analysis 1: Comparison: Sitagliptin and Lansoprazole vs Placebo; Test type: Superiority or Other; p = 0.81, ANCOVA — The p value between treatment groups of C-peptide log (AUC+1) with covariate analysis adjusted for age, sex, baseline C-peptide concentration and duration of diabetes

2. Secondary Outcome: 2 Hour C-peptide AUC in Response to MMTT
Description: Blood samples for C-peptide were collected at baseline (pre-meal) and 15, 30, 60, 90, and 120 minutes post-meal.
Time Frame: Month 6
Population: Of the 70 subjects randomized, 58 completed treatment and analysis.
Measure: Median (95% Confidence Interval); unit: pmol/L
Arm/Group | Sitagliptin and Lansoprazole | Placebo
Number analyzed (Participants) | 40 | 18
pmol/L | 485 [431 to 683] | 675 [495 to 860]
Statistical Analysis 1: Comparison: Sitagliptin and Lansoprazole vs Placebo; Test type: Superiority or Other; p = 0.869, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the August 2010 to May 2013
Groups:
- Sitagliptin and Lansoprazole: Sitagliptin and Lansoprazole: Sitagliptin (dispensed as 50 mg capsules)and Lansoprazole(dispensed as 30 mg capsules) taken for 12 months.
  * Subjects age 11-17 years at Visit 2 will take 1 capsule once daily
  * Subjects age 18-45 years at Visit 2 will take 2 capsules once daily
Arm/Group | Sitagliptin and Lansoprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 2/46 | 1/22
Other Adverse Events (participants affected / at risk) | 44/46 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin and Lansoprazole (N=46) | Placebo (N=22)
Papillary Carcinoma of the Thyroid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin and Lansoprazole (N=46) | Placebo (N=22)
Abdominal Pain (Gastrointestinal disorders) | 11 (15) | 3 (6)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 7 (9)
Nausea (Gastrointestinal disorders) | 8 (8) | 2 (5)
Vomiting (Gastrointestinal disorders) | 10 (10) | 5 (5)
Infections and Infestations-Other (Infections and infestations) | 8 (14) | 2 (2)
Upper Respiratory Infection (Infections and infestations) | 20 (33) | 9 (13)
Neutrophil count decreased (Investigations) | 2 (2) | 3 (5)
Headache (Nervous system disorders) | 15 (16) | 6 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes